CLINICAL TRIAL: NCT00357604
Title: The Effect of the Co-administration of Atazanavir (ATV) and Ritonavir (RTV) on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate in Healthy Female Subjects
Brief Title: Atazanavir and Ritonavir (ATV/RTV) and an Oral Contraceptive in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-285
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV; Protease Inhibitor
MeSH Terms: conditions — HIV Infections | interventions — norgestimate, ethinyl estradiol drug combination; Ethinyl Estradiol; norgestimate; Moxifloxacin; Atazanavir Sulfate; Ritonavir

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Ortho Tri-Cyclen (ethinyl estradiol + norgestimate)
- A2 (Experimental)
  Interventions: Drug: Ortho Tri-Cyclen LO (ethinyl estradiol + norgestimate) + Atazanavir/Ritonavir for 14 days then Ortho Tri-Cyclen for 7 days

INTERVENTIONS:
Drug: Ortho Tri-Cyclen (ethinyl estradiol + norgestimate) — Tablets, Oral, 35 mcg of EE + 0.18/0.215/0.25 mg of NGM, once daily, 28 days.
  Arms: A1
Drug: Ortho Tri-Cyclen LO (ethinyl estradiol + norgestimate) + Atazanavir/Ritonavir for 14 days then Ortho Tri-Cyclen for 7 days — Tablets + Capsules/Capsules, Oral, (25 mcg of EE + 0.18/0.215/0.25 mg of NGM) + 300/100 mg then 35 mcg of EE + 0.18/0.215/0.25 mg of NGM, once daily, 21 days.
  Other Names: Reyataz
  Arms: A2

SUMMARY:
The purpose of this study is to administer a combined oral contraceptive (ethinyl estradiol and norgestimate) with the HIV treatment of atazanavir and ritonavir to healthy females in order to assess if the concentrations of the oral contraceptive change. The safety of this treatment regimen will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential with intact ovarian function who have been on a stable regimen of oral contraceptives for at least 2 months prior to beginning the study
* Documented acceptable Pap smear within 1 year prior to dosing
* Body mass index (BMI) 18-32 kg/m2

Exclusion Criteria:

* Males
* Subjects with an abnormal menstrual cycle during the 2 months prior to the start of the study or during the lead-in period (breakthrough bleeding/spotting)
* History of conditions where the use of oral contraceptives are contraindicated
* Known or suspected carcinoma or suspected estrogen dependent neoplasia
* History of migraine with focal aura
* History of uncontrolled hypertension
* Positive screening test for HIV-1, -2, HIV viral ribonucleic acid (RNA), hepatitis B surface antigen, or hepatitis C antibody

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine the effect of co-administration of atazanavir 300 mg and ritonavir 100 mg on the pharmacokinetics of ethinyl estradiol

SECONDARY OUTCOMES:
To determine the effect of the co-administration of atazanavir 300 mg and ritonavir 100 mg on the pharmacokinetics (PK) of 17-deacetyl norgestimate
To assess the safety of atazanavir 300 mg and ritonavir 100 mg co-administered with the oral contraceptive Ortho Tri-Cyclen LO
To characterize the PK of atazanavir and ritonavir during co-administration with Ortho Tri-Cyclen LO

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Cpu, Inc, San Diego, California, United States